CLINICAL TRIAL: NCT03820791
Title: Using a Visual Poster Communicating Dysphagia-specific Food Procedures as a Complementary Means of Information to Caregivers in Inpatient Care: Usability and Impact
Brief Title: Poster on Dysphagia-specific Food Procedures: Usability and Impact
Acronym: DYSPHAGIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DYSPHAGIA
Record Dates: First submitted 2018-11-15; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poster (Experimental): A poster with pictorial information about dysphagia-specific food procedures placed in patients' rooms for one month
  Interventions: Device: Placement of a poster in patients' rooms
- No poster (No Intervention): No poster is placed in patients' room.

INTERVENTIONS:
Device: Placement of a poster in patients' rooms — Patients and their caregivers will be exposed to the poster for one month
  Arms: Poster

SUMMARY:
The aim of this study is to evaluate the use of a poster containing information on dysphagia-specific food procedures at two levels: utility from the point of view of patients' caregivers, and impact on patients' health. Half the patients will have the poster placed in their room, whereas the other half will not.

DETAILED DESCRIPTION:
Dysphagia is a swallowing disorder that can be associated with clinically relevant complications, and caregivers can play a fundamental role in this process, namely because they feed the patient. However, studies show a lack of professional-caregiver communication in dysphagia, and caregivers' need for more information. Communicating dysphagia-specific food procedures through a visual poster might bridge professional-caregiver communication gaps, with consequences for the patient's health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-acute dysphagia (lesion occurring at least six weeks prior, approximately),
* remaining in inpatient care for at least one month after the first moment of data collection,
* 18 years of age or older,
* receiving regular visits from their family members or caregivers.

Exclusion Criteria:

* Failing to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in patients' aspiration risk before and after placement of the poster in their rooms | 1 month
  Change in patients' risk of aspiration in dysphagia (with the Gugging Swallowing Screen - GUSS)
Change in patients' capacity for oral intake before and after placement of the poster in their rooms | 1 month
  Change in patients' oral intake capacity in dysphagia (with the Functional Oral Intake Scale - FOIS)
Change in patients' oral health before and after placement of the poster in their rooms | 1 month
  Change in patients' oral health in dysphagia (with the Oral Health Assessment Tool - OHAT)
Change in patients' nutritional health before and after placement of the poster in their rooms | 1 month
  Change in patients' nutritional status in dysphagia (with the Mini Nutritional Assessment - MNA)

CONTACTS AND LOCATIONS:
Overall Officials: Irene P Carvalho, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- CINTESIS - Faculty of Medicine of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No